CLINICAL TRIAL: NCT03698825
Title: An Open-label, Multicenter Phase Ib/2a Study of TEW-7197 (Vactosertib) Plus Weekly Paclitaxel As Second-line Treatment for Metastatic Gastric Adenocarcinoma
Brief Title: TEW-7197 with Paclitaxel for the Treatment of Metastatic Gastric Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: MedPacto, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MP-GC-01
Record Dates: First submitted 2018-09-27; First posted 2018-10-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Metastatic Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — vactosertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dose Escalation of TEW-7197 (Experimental): TEW-7191 will be given twice daily (BID) for 5 days followed by 2 days off with a cycle of 4 weeks
  Interventions: Drug: TEW-7197

INTERVENTIONS:
Drug: TEW-7197 — TEW-7197 50mg tablets + Paclitaxel 80 mg/m2 D1, 8, 15 q 4 weeks TEW-7197 dose will be determined through this dose escalation study
  Other Names: vactosertib

SUMMARY:
This is an open-label, single arm study evaluating the safety and tolerability of TEW-7197 in combination with paclitaxel in metastatic gastric cancer patients.

DETAILED DESCRIPTION:
In the dose escalation step (phase 1b), 3 subjects are registered for each dose step, and the DLT is evaluated by administering the investigational product for 1 cycle (28 days). However, for reasons other than toxicity related to the test drug, the patient was given a combination of Paclitaxel and TEW-7197 (Vactosertib) during the DLT evaluation period during the first cycle of the planned TEW-7197.

If more than 80% of the administered dose of (Vactosertib) is not administered, the patient will be considered unevaluable for DLT and another patient will be enrolled. At the end of one cycle of each cohort, the SMC decides whether to proceed to the next cohort. After completing the DLT evaluation of the final phase 1 cohort, the recommended dose to proceed in the dose expansion phase (Phase 2a) is determined. For subjects who have completed one cycle (DLT evaluation period), administer the investigational drug at the same dose until disease progression or unacceptable toxicity occurs. Tumor imaging (CT or MRI) for tumor evaluation is performed after screening and C1D1. Assessment every 6 weeks (±2 weeks) and at the end of treatment (EOT/DC). As efficacy evaluation items, PFS, OS, ORR, and DCR are evaluated according to RECIST 1.1, and the amount of change in the biomarker is confirmed.

In the dose expansion phase (phase 2a), 50 patients will be enrolled at the dose determined in the dose escalation phase. Tumor imaging (CT or MRI) for tumor evaluation is evaluated every 6 weeks (±2 weeks) after screening and C1D1, and at the end of treatment (EOT/DC). As validity evaluation items, PFS, OS, ORR, and DCR according to RECIST 1.1 are evaluated, and the amount of change in the biomarker is confirmed.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women over 19 years of age
2. Patients diagnosed with histologically or cytologically metastatic gastric cancer
3. Patients corresponding to ECOG Performance Status 0
4. The 5-Fluorouracil family (5-Fluorouracil) is the primary treatment for metastatic gastric cancer.

   Patients who received additional Trastuzumab coalescing therapy for Cisplatin (Oxaliplatin) and Platinum (Oxaliplatin) or HER2-positive.
5. Patients with evalable lesions according to Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST 1.1)
6. Patients with the following laboratory test values during screening:

   * Bilirubin is not more than 1.5 times the upper limit of normal (ULN)
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) not more than 3 times ULN (if liver metastasis, not more than 5 times ULN)
   * Serum cretin is not more than 1.5 times the ULN
   * Absolute neutrophil count (ANC)가 1,000 cells/µL 이상
   * Platelet count is over 80,000/µL
   * Hemoglobin count 가 9.0 g/dL 이상
7. Patients who voluntarily agreed to participate in the clinical trial after hearing the explanation of this clinical trial.

Exclusion Criteria:

1. Patients with unresolved chronic toxicity of CTC grade 2 or higher in previous chemotherapy
2. Patients who have received chemotherapy or chemotherapy within two weeks prior to screening
3. Patients who have undergone major surgery or radiation treatment within four weeks prior to screening
4. Patients who have received medication for other clinical trials before screening and have less than 5 times the period of this half-life. Patients who are less than two weeks from the date of final administration if the half-life of the previous clinical trial drug is not clear.
5. Patients previously treated with paclitaxel
6. Patients who previously received treatment targeting the TGF-£ signaling pathway
7. Patients who cannot take tablets
8. Patients who are neurologically unstable due to overall metastasis in the central nervous system or who have increased the amount of steroid to alleviate the central nervous system signs within two weeks before screening.
9. If another type of tumor is present, or within three years prior to screening, another tumor is present.

   diagnosed patients (except for single basal cell carcinoma, thyroid cancer and cervical cancer-insitu)
10. Patients with a history of congestive heart failure or myocardial infarction that is not controlled by medication
11. Pregnant women who are positive for pregnancy test results in this clinical trial and contraception by themselves and their partners during the safety follow-up period after treatment (e.g., infertility surgery, intrauterine, oral contraceptives, liver wall contraception, and other hormone delivery systems, creams, jellies, etc.)
12. Patients with evidence of cirrhosis above Child-Pugh B or C. For HBV or HCV-linked chronic hepatitis or cirrhosis Child-Pugh A, it can be registered for clinical trials if the liver function is reliably maintained through medication.
13. Other patients who are deemed unfit to participate in the study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2022-01-03 (Actual); Study Completion 2022-12-28 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 4 weeks
  To define the MTD and determine RP2D

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events assessed by NCI CTCAE v5.0 | from screening through study completion (up to 28 days after the last dose of TEW-7197), an average of 1 year.
  To evaluate safety profile of TEW-7197 with regards to frequency, type, grade, and seriousness, and causality of treatment-related clinical and laboratory adverse events including, but not limited to, AST, ALT, total bilirubin, serum creatinine, etc.
Overall survival | every 2 cycles (8 weeks) and end-of-treatment (EOT) time point. EOT is defined as within 7 days from the last dose of study medication by the protocol.
  Overall survival (months, median) defined by RECIST 1.1
Objective response | every 2 cycles (8 weeks) and end-of-treatment (EOT) time point. EOT is defined as within 7 days from the last dose of study medication by the protocol.
  Objective response rate (%) defined by RECIST 1.1
pharmacokinetics of TEW-7197 | At cycle 1 (each cycle is 28 days)
  Peak Plasma Concentration (Cmax) of TEW-7197 Area under the plasma concentration versus time curve (AUC) of TEW-7197

OTHER OUTCOMES:
pSMAD as a pharmacodynamic marker | At baseline and cycle 1 (each cycle is 28 days)
  pSMAD in peripheral blood mononuclear cell determined by immunohistochemistry

CONTACTS AND LOCATIONS:
Overall Officials: Sunjin Hwang, MD, Study Director — MedPacto, Inc.
Locations (6):
- South Korea (6):
  - Hallym University Medical Center, Anyang-si
  - Hwasun Chunnam university hospital, Hwasun
  - Chung-Ang University hospital, Seoul
  - Gangbuk Samsung Medical Center, Seoul
  - Gangnam Severance, Seoul
  - Shinchon Severance, Seoul

IPD SHARING:
Plan to Share IPD: No